CLINICAL TRIAL: NCT03359811
Title: Four Quadrants Transverse Abdominus Plane (4Q-TAP) Block With Plain and Liposomal Bupivacaine vs. Thoracic Epidermal Analgesia (TEA) in Patients Undergoing Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC) on an Enhanced Recovery Pathway: A Non-inferiority Randomized Controlled Trial
Brief Title: Four Quadrants Transverse Abdominus Plane (4Q-TAP) Block With Plain and Liposomal Bupivacaine vs. Thoracic Epidermal Analgesia (TEA) in Patients Undergoing Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC) on an Enhanced Recovery Pathway
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0492; NCI-2018-00999 (Other: NCI)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Peritoneal Cancer
Keywords: Local Anesthetic Solution; Bupivacaine HCl; Liposomal Bupivacaine; Peritoneal Cancer
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-of-Care Thoracic Epidural Analgesia (TEA) (Experimental): An epidural catheter placed before induction of anesthesia by an anesthesiologist. A bolus or infusion of the local anesthetic solution with or without the addition opioids given before surgical incision according to anesthesia provider's clinical judgment.
  Interventions: Drug: Local Anesthetic Solution
- 4Q-TAP Blocks (Active Comparator): Participants have an ultrasound guided 4Q-TAP block. A maximum of 80 cc of a solution consisting of 30 mg of bupivacaine HCl in 10 cc of preservative free normal saline (PFNS) and 65 mg of liposomal bupivacaine in 10 cc of PFNS injected before surgical incision in each of the four quadrants.
  Interventions: Drug: Bupivacaine HCl; Drug: Liposomal Bupivacaine

INTERVENTIONS:
Drug: Local Anesthetic Solution — A bolus or infusion of local anesthetic solution with or without the addition opioids given before surgical incision according to anesthesia provider's clinical judgment.
  Arms: Standard-of-Care Thoracic Epidural Analgesia (TEA)
Drug: Bupivacaine HCl — 30 mg of Bupivacaine HCl in 10 cc of preservative free normal saline (PFNS) injected before surgical incision in each of the four quadrants.
  Arms: 4Q-TAP Blocks
Drug: Liposomal Bupivacaine — 65 mg of Liposomal Bupivacaine in 10 cc of PFNS injected before surgical incision in each of the four quadrants.
  Other Names: EXPAREL
  Arms: 4Q-TAP Blocks

SUMMARY:
The goal of this clinical research study is to compare the effects of 4 quadrant TAP block (4Q-TAP block) with the standard-of-care thoracic epidural analgesia (TEA) in patients recovering from cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS-HIPEC).

A 4Q-TAP block is also known as an abdominal wall block and TEA is also known as a thoracic epidural. Both are types of anesthetics but are given in different ways. A 4Q-TAP block is when anesthetic injections are given in 4 different parts of the abdomen. A TEA is when an anesthetic injection is given in the space surrounding the spinal cord through your back.

This is an investigational study. The surgery and the levels of anesthetic participant is receiving are standard-of-care. It is investigational to compare 4Q-TAP block with TEA.

Up to 140 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Baseline Tests:

If participant agrees to take part in this study, within 60 days before participant's surgery:

* Participant will have a physical exam.
* Blood (about 8 teaspoons) will be drawn for routine tests.
* Participant will complete a questionnaire about the quality of recovery. Participant's responses before surgery will be compared to participant's responses after surgery. It should take about 5 minutes to complete.

Study Groups/Procedures:

Participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups on the morning of participant's surgery. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If participant is in Group 1, participant will receive standard-of-care TEA before participant goes to sleep.
* If participant is in Group 2, participant will receive the 4Q-TAP block injections after participant is asleep.

If participant is in Group 1, participant will have a catheter placed in participant's back before surgery so that the TEA can be infused. If needed, participant may receive an injection of numbing medication and/or pain medication before the catheter is placed. Participant will sign a separate consent for the placement of the catheter.

If participant is in Group 2, participant will receive up to four (4) injections of 4Q-TAP block directly into different parts of the abdomen. These injections will take place after participant has been given general anesthesia. An ultrasound will be used to guide these injections. Participant will not be awake for these injections.

Both groups will sign a separate consent for the surgery that explains the procedures and the risks. Participant may receive standard drugs during surgery. The study staff can tell participant about the risks of these drugs and how they are given.

For both groups, information about the surgery will be collected while participant is in the operating room.

Post-Surgery:

After surgery, participant will receive standard drugs for pain as needed. Participant will be asked to complete a questionnaire about the quality of participant's recovery on the following days after surgery:

* Days 1-3
* Day 5
* Day 7
* Day 10 and
* Day 30

The questionnaire should take about 5 minutes each time. Participant will complete the questionnaire in person or participant will be called on the phone to complete it if participant has already left the hospital.

On Days 1, 2, and 7 after surgery, blood (about 8 teaspoons each time) will be drawn for routine tests.

After participant leaves the hospital, researchers will collect information from participant's medical record about participant's standard follow-up visits.

Length of Study Participation:

Active participation in this study will be complete 30 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed consent
2. 18 years old or older
3. American Society of Anesthesiologists physical status (ASA) 1-3
4. Scheduled surgery: open elective CRS-HIPEC
5. Able to complete the QoR 15 questionnaire
6. Patients scheduled to receive intraoperative chemotherapy

Exclusion Criteria:

1. Thrombocytopenia (platelet count: <100,000 cell/dL), coagulopathy (International Normalized Ratio > 1.5, PT>16.5 seconds or aPTT > 35.9 seconds)
2. Bupivacaine or liposomal bupivacaine sensitive or known allergy;
3. Pregnancy or breastfeeding patients
4. Patients with recent (within 60 days preoperatively) history severe hepatic disease (defined as liver injury with encephalopathy plus impaired synthetic liver function (i.e. >1.5)
5. Patients with recent (within 15 days preoperatively) history deteriorate kidney function (creatinine serum concentrations > 2.5 mg/dL or eGFR < 30 mL/kg/min)
6. Chronic opioid use defined as daily opioid use for more than one month prior the scheduled date of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from November 2017 to February 2020.
Pre-assignment Details: A total of 75 participants consented, 5 participants were inevaluable.
Groups:
- Standard-of-Care Thoracic Epidural Analgesia (TEA): Participants allocated to the TEA group had an epidural catheter placed before induction of anesthesia. The catheter was placed between the thoracic vertebral spaces 8 and 12 according to standard procedure. A bolus or infusion of local anesthetic solution with or without the addition opioids (bupivacaine 0.075% ± hydromorphone 2-5 mcg/mL or bupivacaine 0.075% ± fentanyl 5 mcg/mL, basal rate 8 mL/h, bolus 3 mL every 10 min) were given before surgical incision according to the anesthesiologist's clinical judgment. If deemed appropriate, a precision epidural bolus of hydromorphone (300-800 micrograms) was administered.
- Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block: Participants in 4Q-TAP group received maximum of 80. cc of a solution consisting of 150 mg of bupivacaine HCl and 266 mg of liposomal bupivacaine divided between each of the four quadrants after induction of anesthesia. All 4Q-TAP were done after induction of general anesthesia and under ultrasound guidance.
Period: Overall Study
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Started | 35 | 35
Completed | 33 | 35
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics data is only available for the participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 29 | 53
  >=65 years | 9 | 6 | 15
Age, Continuous [Median (Full Range); unit: years] | 58 [20 to 74] | 57 [25 to 72] | 58 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 15 | 14 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 68
Median BMI [Median (Full Range); unit: kg/m^2] | 26.6 [16.5 to 47.9] | 25.4 [19.3 to 51.3] | 26.6 [16.5 to 51.3]
History of Depression [Count of Participants; unit: Participants]
  No | 27 | 27 | 54
  Yes | 6 | 8 | 14
Preoperative antidepressants [Count of Participants; unit: Participants]
  No | 27 | 28 | 55
  Yes | 6 | 7 | 13
Preoperative Opioids [Count of Participants; unit: Participants]
  No | 32 | 34 | 66
  Yes | 1 | 1 | 2
Median Anesthesia Duration [Median (Full Range); unit: Minutes] | 649 [216 to 935] | 634 [257 to 1017] | 641 [216 to 1017]
Volatile anesthesia [Count of Participants; unit: Participants]
  No | 3 | 5 | 8
  Yes | 30 | 30 | 60
Median propofol consumption [Median (Full Range); unit: milligrams] | 672.7 [140 to 3288] | 200 [2.3 to 12234.3] | 235 [2.3 to 12234.3]
Dexmedetomidine use [Count of Participants; unit: Participants]
  No | 4 | 4 | 8
  Yes | 29 | 31 | 60
Median Crystalloids use [Median (Full Range); unit: mililiters] | 3000 [1000 to 6400] | 3050 [1000 to 5800] | 3050 [1000 to 6400]
Red blood cell transfusion intraoperatively [Count of Participants; unit: Participants]
  No | 32 | 33 | 65
  Yes | 1 | 2 | 3
Frozen plasma transfusions intraoperatively [Count of Participants; unit: Participants]
  No | 33 | 34 | 67
  Yes | 0 | 1 | 1
Perfusion completed [Count of Participants; unit: Participants]
  No | 4 | 4 | 8
  Yes | 29 | 31 | 60
Urinary output [Median (Full Range); unit: mililiters] | 665 [180 to 2370] | 900 [30 to 2225] | 783 [30 to 2370]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of TEA vs 4Q-TAP in QoR at Postoperative Day (POD)2
Description: To compare the efficacy of 4 quadrants TAP blocks (4Q-TAP) versus Thoracic Epidural Analgesia (routine care) on the quality of recovery 48 hours after CRS-HIPEC surgery, measure by QoR-15 changes from Pre-Op to POD2. The QoR scale is a validated scoring system that allows for the quantification of a patient's early postoperative health status. The minimum score 0 and maximum score 150. The higher score mean a better outcome.
Time Frame: 48 hours after CRS-HIPEC surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
score on a scale | -45 [-89 to 0] | -50 [-88 to 23]

2. Secondary Outcome: 4Q-TAP Versus TEA on Postoperative Pain
Description: Pain intensity at rest and cough measure using a Validity and Reliability of the Verbal Numerical Rating Scale (VNRS) (0 = no pain - 10 = worst pain ever). Higher numerical scores on the scale indicate more pain, thus a worse outcome. Data reported as time-weighted pain scores from discharge from the PACU until 48 hours after the end of surgery.
Time Frame: 48 hours after CRS-HIPEC surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
score on a scale
  Pain at Rest | 3 [0 to 10] | 4 [0 to 10]
  Pain with Cough | 5 [1 to 10] | 5 [1 to 10]

3. Secondary Outcome: Comparison of the Total Opioid Consumption Between Patients With 4Q-TAP Versus TEA
Description: Opioid Consumption reported as morphine equivalents required during the 48 hours after the end of surgery.
Time Frame: During the 48 hours after CRS-HIPEC surgery
Measure: Median (Full Range); unit: morphine milligram equivalents (MME)
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
morphine milligram equivalents (MME) | 4.5 [0 to 51] | 21 [1.8 to 108.8]

4. Secondary Outcome: Comparison of the Length of Stay (LOS) Between Patients With 4Q-TAP Versus TEA
Description: Length of stay calculated from day of surgery to date of hospital discharge.
Time Frame: Length of stay calculated from day of surgery to date of hospital discharge, up to 46 days
Measure: Median (Full Range); unit: days
Groups:
- 4Q-TAP Blocks: Participants in 4Q-TAP group received maximum of 80. cc of a solution consisting of 150 mg of bupivacaine HCl and 266 mg of liposomal bupivacaine divided between each of the four quadrants after induction of anesthesia. All 4Q-TAP were done after induction of general anesthesia and under ultrasound guidance.
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | 4Q-TAP Blocks
Number analyzed (Participants) | 33 | 35
days | 11 [4 to 24] | 11 [4 to 46]

5. Secondary Outcome: Number of Participants With Adverse Events Related to 4Q-TAP Versus TEA
Description: An adverse event is any symptom, sign, illness, or experience which develops or worsens during the course of the study, whether or not the event is considered related to study drug. Adverse events (AEs) related to the study interventions recorded within the first 48 hours after the end of surgery.
Time Frame: 48 hours after CRS-HIPEC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
Participants | 3 | 1

6. Secondary Outcome: Number of Participants With Incidence of Opioid-Related Adverse Events Related to 4Q-TAP Versus TEA 48
Description: Opioid-related adverse (i.e. respiratory depression, pruritus, sedation, delirium) within the first 48 hours after the end of surgery.
Time Frame: Within the first 48 hours after the end of CRS-HIPEC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
Participants | 7 | 7

7. Secondary Outcome: Number of Participants With Incidence of Postoperative Complications and Morbidity in Patients Receiving 4Q-TAP Versus TEA
Description: Postoperative complications recorded using Clavien-Dindo scale and POMS.
Time Frame: 48 hours after CRS-HIPEC surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
Number analyzed (Participants) | 33 | 35
Participants
  Pulmonary Complications | 5 | 8
  Renal Complications | 5 | 5
  Gastrointestinal Complications | 1 | 0
  Cardiac Complications | 7 | 4
  Hematological Complications | 2 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected within the first 48 hours after end of surgery, up to 30 days
Arm/Group | Standard-of-Care Thoracic Epidural Analgesia (TEA) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/35
Other Adverse Events (participants affected / at risk) | 17/33 | 16/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard-of-Care Thoracic Epidural Analgesia (TEA) (N=33) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block (N=35)
Intraabdominal Abscess (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard-of-Care Thoracic Epidural Analgesia (TEA) (N=33) | Four Quadrant Transverse Abdominus Plane (4Q-TAP) Block (N=35)
Dry mouth (Gastrointestinal disorders) | 2 | 4
Hypotension (Cardiac disorders) | 14 | 8
Ileus (Gastrointestinal disorders) | 1 | 0
Low urinary input (Renal and urinary disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 17 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Sedation (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03359811/Prot_SAP_000.pdf